CLINICAL TRIAL: NCT06973824
Title: A Twenty-years' Experience in Pituitary Disease: Identification of Prognostic Factors in Pituitary Tumors
Brief Title: A Twenty-years' Experience in Pituitary Disease.
Acronym: TYEPDD
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Doglietto Francesco, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6546
Record Dates: First submitted 2025-01-22; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Pituitary Adenoma; Pituitary Cancer; Pituitary Disease
MeSH Terms: conditions — Pituitary Neoplasms; Pituitary Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with pituitary tumors: Patients with pituitary tumors, underwent surgical resection
  Interventions: Other: Frequency of disease recurrence

INTERVENTIONS:
Other: Frequency of disease recurrence — To collect data of pituitary disease recurrence

SUMMARY:
Pituitary tumors represent a heterogeneous group of neoplasms by histotype. The pituitary adenomas are the most frequent heteroformation, among those affecting the pituitary gland, followed by meningiomas, craniopharyngiomas, germosomes and tumours secondary, such as metastases and lymphomas. Since these conditions are considered rare, the data epidemiology and prognosis to predict the natural history of these diseases can not be considered conclusive. Pituitary adenomas are a useful model for epidemiology in the study of pathology pituitary. Over the past 20 years, several attempts have been made to identify unique prognostic factors, which predict the outcome of these pathologies, but without To arrive at a definitive classification. The purpose of this study aims to collect clinical, biochemical, morphological and pathological data on the retrospective and prospective cohort of over 1600 patients undergoing neurosurgical removal of pituitary tumors in the last 20 years, to develop a prognostic classification.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent surgery for pituitary tumors;
* pathology diagnosis of pituitary tumors;
* patients older then 18 years at diagnosis of pituitary tumors;
* 2 years follow-up;

Exclusion Criteria:

* age lower then 18 years
* follow-up shorter than 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older then 18 years with diagnosis of pituitary tumors (pituitary adenoma, pituitary neuroendocrine tumors, meningiomas, craniopharingiomas, germinoma, metastasis)
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2028-02-15 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Tumor recurrence | From enrollement to last observation at 24 months of follow-up
  Frequency of tumor recurrence at 24 months of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Doglietto, Prof, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Rome, IT, Italy

IPD SHARING:
Plan to Share IPD: Undecided